CLINICAL TRIAL: NCT06009471
Title: A Multicenter Clinical Study of rTMS for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCYJ-B06
Record Dates: First submitted 2023-06-25; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; repetitive transcranial magnetic stimulation(rTMS); Unified Parkinson's Disease Rating Scale (UPDRS); Montreal Cognitive Assessment Scale (MoCA); activity of daily living(ADL); PD Sleep Scale (PDSS); King's Parkinson's Pain Assessment (KPPS)
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: A total of 200 patients with Parkinson's disease were enrolled in each center and randomly divided into control group (routine treatment) and observation group (routine treatment +rTMS).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): All participants were treated with routine treatment in Neurology.
  Interventions: Other: Routine treatment in Neurology
- Experimental group (Experimental): All participants were treated with routine treatment in Neurology and rTMS treatment.
  rTMS parameters were set to stimulate the site: bilateral primary motor cortex; Stimulus frequency :5Hz; Pulse number: 1000 pulses per day, 500 on the left and 500 on the right; Stimulus intensity :90% resting threshold; Coil: 70mm round coil; Once a day, 30 minutes each time, 5 days a week for 4 weeks
  Interventions: Device: Routine treatment in Neurology and rTMS

INTERVENTIONS:
Other: Routine treatment in Neurology — Routine treatment in Neurology department, including drug treatment,etc.
  Arms: Control group
Device: Routine treatment in Neurology and rTMS — Add rTMS to routine treatment. Low frequency rTMS is often used to treat cortical hyperexcitability and high frequency rTMS to treat hypoexcitability
  Arms: Experimental group

SUMMARY:
Through rTMS, motor dysfunction and non-motor dysfunction of PD patients can be improved, working and living ability and quality of life of patients can be improved, and social burden and family burden can be reduced.

DETAILED DESCRIPTION:
According to the inclusion criteria, a total of 200 patients with Parkinson's disease were planned to be enrolled in each center, and randomly divided into control group (conventional treatment) and observation group (conventional treatment +rTMS) for a treatment cycle of 4 weeks. They were followed up for 3 months before treatment, 2 weeks and 4 weeks, respectively, after treatment, to evaluate the efficacy and function. The unified Parkinson's Disease Rating Scale (UPDRS) was used. Cognitive function assessment Monteller Cognitive Assessment Scale (MoCA); Barthel Index for daily living activities; Depression assessment Hamilton Depression Scale (HAMD); Hamilton Anxiety Scale (HAMA); Sleep assessment PD Sleep Scale (PDSS); Pain assessment King Parkinson's Pain Assessment (KPPS) and adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn-YAHR classification is between 1 and 2；
* Have a primary school education or above and can read the scale used in this study;
* MoCA score between 20 and 24, mild cognitive impairment ;
* Aged between 30 and 80, regardless of gender；
* Voluntarily participate and sign informed consent.

Exclusion Criteria:

* patients with cerebrovascular accident, craniocerebral injury and other diseases affecting muscle tension;
* patients with serious mental disorders and cognitive disorders who cannot cooperate with assessment;
* patients with severe liver, kidney, heart dysfunction and severe physical disorders;
* Implanted devices such as pacemakers are installed inside the body;
* drug-induced Parkinson's syndrome or Parkinson's superposition syndrome;
* Have a history of epilepsy;
* Women during pregnancy and breastfeeding.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's disease rating Scale （UPDRS） | The assessments are conducted at the baseline, 2nd week, 4th week, and 3 months after the end of treatment.
  16 items, each with a score of 0-4, and the score is directly proportional to the severity of PD motor symptoms.
Montreal Cognitive Assessment Scale (MoCA) | The assessments are conducted at the baseline, 2nd week, 4th week, and 3 months after the end of treatment.
  Full score of 30 points,>=26 points normal,. Mild cognitive impairment (MCI) on a scale of 18-26, moderate on a scale of 10-17, and severe on a scale of<10.
King's Parkinson's Pain Assessment (KPPS) | The assessments are conducted at the baseline, 2nd week, 4th week, and 3 months after the end of treatment.
  Evaluate the pain degree and quality of life of patients with Parkinson's disease, including 14 items in 7 aspects, including skeletal muscle pain, Chronic pain, symptom fluctuation related pain, nocturnal pain, orofacial pain, distention pain, and nerve root pain. Each score is expressed as pain severity (0-3 levels) multiplied by frequency (0-4 levels), that is, 0-12 points. The total score is 168 points. The higher the score, the more severe the pain.
PD Sleep Scale (PDSS) | The assessments are conducted at the baseline, 2nd week, 4th week, and 3 months after the end of treatment.
  Evaluate the patient's sleep status, with a total of 15 items on the scale. Each item is scored on a scale of 0-10 points, with a lower score indicating poorer sleep status.
Activities of daily living Assessment - Barthel | The assessments are conducted at the baseline, 2nd week, 4th week, and 3 months after the end of treatment.
  The total score of the index is 100 points, and the higher the score, the better the self-care ability and the less dependence. Those scoring above 60 can basically complete basic Activities of daily living, 59-41 need some help to complete, 40-21 need a lot of help. Those who score below 20 are in complete need of help and cannot take care of themselves.

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAMD) | The assessments are conducted at the baseline, 2nd week, 4th week, and 3 months after the end of treatment.
  Evaluate depressive status, including 14 5-level scoring items (0-4 points) and 10 3-level scoring items (0-2 points). Score<8, no depression; 8 to 35 points, may be mild or moderate depression 35 points, may be severe depression.
Hamilton Anxiety Scale (HAMA) | The assessments are conducted at the baseline, 2nd week, 4th week, and 3 months after the end of treatment.
  Include 14 projects. All items of HAMA adopt a 5-level scoring method of 0~4 points, and the criteria of each level are: (0) is Asymptomatic; (1) Light; (2) Moderate; (3) Heavy; (4) Extremely heavy. The total score of HAMA can better reflect the severity of anxiety symptoms. The total score can be used to evaluate the severity of anxiety symptoms and evaluate the effectiveness of various drugs and psychological interventions in patients with anxiety and depression disorders. According to the data provided by the collaborative group of the Chinese scale, if the total score exceeds 29 points, it may be severe anxiety; Above 21 points, there must be obvious anxiety; If the score exceeds 14, there must be anxiety; If the score exceeds 7, there may be anxiety; If the score is less than 7, there are no symptoms of anxiety. Generally speaking, the total score of HAMA is higher than 14 points, indicating clinically significant anxiety symptoms for the evaluated subject.

CONTACTS AND LOCATIONS:
Locations (1):
- rTMS, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No